CLINICAL TRIAL: NCT06627452
Title: The Effectiveness of Dynamic Neuromuscular Stabilization on Incontinence Severity, Pelvic Floor Muscle Strength and Quality of Life in Women With Urinary Incontinence
Brief Title: Effectiveness of DNS on Incontinence Severity, Pelvic Floor Strength and QoL in Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Assoc. Prof., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: _IstanbulUCdılanacar13579.....
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2024-09

CONDITIONS: Urinary Incontinence , Stress; Urinary Incontinence (UI); Exercise
Keywords: dynamic neuromuscular stabilization; kegel exercise; urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): Participants in Dynamic Neuromuscular Stabilization(DNS) will perform exercises with a physiotherapist twice a week and at home three days a week. The sessions will last approximately 30 minutes and will be conducted five days a week for 12 weeks.
  Interventions: Other: Dynamic Neuromuscular Stabilization Training
- Control Group (Active Comparator): Participants in Pelvic Floor Muscle Training (PFMT) will be taught pelvic floor exercises through vaginal palpation. They will perform the exercises with a physiotherapist two days a week and at home three days a week. The sessions will last approximately 30 minutes and will be conducted five days a week for 12 weeks.
  Interventions: Other: Pelvic Floor Muscle Training

INTERVENTIONS:
Other: Dynamic Neuromuscular Stabilization Training — Patients will be taught how to perform exercises in different developmental positions both manually and verbally by the DNS therapist. In the DNS concept, proper breathing patterns are important alongside stabilization, and elastic bands will be used to regulate intra-abdominal pressure (IAP) and teach correct breathing. The elastic band will be secured around the chest just below the ribcage, and the patient will be asked to expand the elastic band in all directions while inhaling, thereby regulating the IAP. After teaching IAP guidance, exercises will be conducted in developmental positions with IAP regulation. The exercises will be conducted twice a week under the supervision of a physiotherapist, and three days at home, with sessions lasting approximately 30 minutes, for a total of five days a week over a period of 12 weeks.
  Arms: Study Group
Other: Pelvic Floor Muscle Training — Pelvic floor exercises involving both slow and fast muscle contractions will be taught to patients through vaginal palpation. During fast contractions, patients will be instructed to quickly contract and relax their pelvic floor muscles. During slow contractions, patients will be asked to gradually squeeze their pelvic floor muscles, hold for 10 seconds, and then slowly relax. Each set of pelvic floor exercises will consist of 10 fast contractions and 10 slow contractions. Patients will perform pelvic floor exercises twice a week with a physiotherapist and three days at home. The exercises will be done in sets throughout the day, lasting approximately 30 minutes, and will be conducted over a period of 12 weeks.
  Arms: Control Group

SUMMARY:
The aim of this study is to investigate the effects of Dynamic Neuromuscular Stabilization (DNS) Training on incontinence severity, pelvic floor muscle strength, and quality of life in women with Urinary Incontinence, compared to Pelvic Floor Muscle Training (PFMT). The hypothesis of the study is that DNS Training will be at least as effective as PFMT in terms of its impact on incontinence severity, pelvic floor muscle strength, and quality of life in women with Urinary Incontinence. A total of 56 women diagnosed with urinary incontinence will be included in the study. Participants will be divided into two groups: DNS and PFMT, and will engage in the designated exercise program 5 days a week for a total of 12 weeks. All participants will undergo an initial assessment before starting treatment, and a final assessment will be conducted by the same physiotherapist after the treatment.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is defined by the International Continence Society as involuntary leakage of urine and is a symptom that can objectively be demonstrated, leading to social and hygienic problems. UI negatively affects daily life activities, perception of health status, and mental and social well-being, thereby reducing individuals; health-related quality of life. UI is commonly observed in women, with a reported prevalence ranging from 25% to 45%. There are three main types of urinary incontinence: stress urinary incontinence, urge urinary incontinence, and mixed urinary incontinence. The most commonly seen type, stress urinary incontinence, is defined as involuntary urine leakage due to a sudden increase in intra-abdominal pressure (IAP) during activities such as coughing, sneezing, exertion, or physical activity without detrusor contraction. It generally occurs after childbirth or during pregnancy. Risk factors for stress urinary incontinence in women include a higher number of births, age, smoking, lung disease, and obesity. One of the significant causes of UI is the weakness of the pelvic floor muscles (PFM).

It is known that the PFM helps stabilize the bladder neck and contributes to continence control by increasing intraurethral pressure. The PFM also aids in stabilizing the lumbopelvic region (core). Studies show that the transverse abdominis (TrA), one of the most essential muscles providing core stabilization, works synergistically with the PFM. This co-activation has been reported to enhance pelvic stability and support urinary control, modulating IAP and load transfer. In this context, in addition to PFM training, stabilization exercises have begun to be included in treatment programs for patients with UI as a first-line treatment.

Dynamic Neuromuscular Stabilization (DNS) is a neuromuscular and functional stabilization approach based on developmental kinesiology models, utilizing the normal motor development process to assess and treat motor disorders. The primary aim is to restore the physiological movement patterns defined by developmental kinesiology. DNS provides stabilization of the spine and surrounding muscles during static and dynamic movements. Deep spinal flexors and extensors, multifidus, diaphragm, pelvic floor muscles, and abdominal muscles are part of this system. The co-contractions of these muscles increase IAP, thereby aiding. This also helps with stabilization. DNS is based on the principle that the core muscle system works synergistically with various components. When part of this system is weak or dysfunctional, it can also affect the functioning of other core muscles. DNS exercises focus on comprehensive activation and strengthening of the entire core muscle system rather than targeting individual muscles one by one. In this context, DNS training includes the development of pelvic floor muscles along with the improvement of core (lumbopelvic) stabilization.

It is known that the strength of the pelvic floor muscles (PFM) decreases in women with UI, and strengthening these muscles plays a crucial role in controlling incontinence. However, there are also studies reporting low stabilization in women with UI. Considering that stress urinary incontinence occurs due to a sudden increase in intra-abdominal pressure during physical activity, regulating IAP and improving stabilization could be more effective in controlling UI. The DNS method, which targets lumbopelvic stabilization along with PFM training and focuses on intra-abdominal pressure regulation, has been shown to have positive effects on various neuromuscular disorders and postural dysfunctions. There is only one pilot study in the literature investigating the effects of DNS training on women with UI. This study reported that DNS improved PFM strength more than Kegel exercises. Given this information, it is hypothesized that DNS training may more effectively reduce the severity of urinary incontinence in women compared to PFM training. Therefore, this research aims to compare the effects of DNS training on urinary incontinence severity in women with urinary incontinence to PFM training.

METHOD

The research will include young adult women who have been diagnosed with urinary incontinence and volunteered to participate. Participants will be divided into two parallel groups (1:1): the dynamic neuromuscular stabilization (DNS) group and the pelvic floor muscle training (PFMT) group. Our study will be conducted per the Helsinki Declaration, and all participants will be informed about the research and provide written consent.

Indıviduals will be randomly divided into the dynamic neuromuscular stabilization (DNS) and pelvic floor muscle training (PFMT) groups. The treatment program will be implemented by the same experienced physiotherapist, who holds a training certificate in both DNS and PFMT. Participants will be taught how to perform the exercises correctly and receive an exercise sheet containing exercises to perform at home as a guide.

Dynamic Neuromuscular Stabilization Training Participants in this group will undergo Dynamic Neuromuscular Stabilization exercises. The exercises will be performed with the physiotherapist twice a week, while participants will practice at home three days a week, with each session lasting approximately 30 minutes. This program will continue for 12 weeks, totaling five days of exercise per week. The DNS therapist will manually and verbally instruct the participants on how to perform exercises in various developmental positions.

Pelvic Floor Muscle Training Pelvic floor exercises will be taught to patients through vaginal palpation. The exercises will be performed with the physiotherapist twice a week, while participants will practice at home three days a week. To increase adherence to the home exercises and encourage proper execution, a PTKE schedule and a document demonstrating and explaining the pelvic floor exercises will be provided. Exercise schedules will be checked weekly.

Patients will be instructed to perform pelvic floor exercises in sets for approximately 30 minutes daily over a period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severity stress urinary incontinence based on symptoms
* Being literate
* Aged between 18 and 65
* Not having received any conservative treatment in the last 6 months.

Exclusion Criteria:

* Presence of prolapse
* Diagnosis of overactive bladder
* Ongoing urinary tract infection
* Use of medication for urinary incontinence
* Pregnancy
* Lack of cooperation for assessment and/or treatment
* Having undergone uro-surgical procedures within the last two years
* Patients with serious systemic diseases that would prevent them from exercising (such as cardiovascular disease, COPD, stroke, and/or cancer, etc.)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Incontinence Severity Index (ISI) | 12 WEEKS
  Patients incontinence severity will be assessed using the Incontinence Severity Index (ISI). The index has two questions: 1) How often do you leak urine? (0=Never, 1=Less than once a month, 2=Once a month, 3=Several times a week, 4=Almost every day/night), and 2) How much urine do you leak? (0=None, 1=A few drops, 2=Small spots, 3=More). The result obtained from this index is the product of the two items that assess the frequency and amount of incontinence.
  The total score ranges from 1 to 12 and is categorized into four levels of incontinence severity: Mild (1 and 2 points), Moderate (3, 4, and 6 points), severe (8 and 9 points), and very severe (12 points).
24-Hour Pad Test | 12 WEEKS
  The pad test is one of the assessments that provide information about the severity of incontinence. One day before the examination, patients will be instructed to place a dry pad in their underwear after their first morning urination and continue their daily activities. They should change the pad every 4 to 6 hours to prevent evaporation and store the used pads in a sealed bag.
  Patients must bring all pads used until the next morning, along with a dry pad sample, for examination. The pads will be weighed on a sensitive scale to calculate the amount of urinary leakage. In the 24-hour pad test, values above 4 grams are considered significant, with incontinence severity classified as mild (≥4-20 grams/24 hours), moderate (21-74 grams/24 hours), and severe (≥75 grams/24 hours).
Urinary Diary | 12 WEEKS
  A urinary diary is an assessment tool that records the frequency of urination, types and amounts of fluids consumed, and the frequency and severity of incontinence over a specified period. The recommended duration for keeping the diary is typically 1 to 7 days. A 3-day diary has been noted as an appropriate outcome measure for clinical studies evaluating stress incontinence treatments.
  Patients are advised not to change their usual urination habits or fluid intake while completing the diaries. A total of three diaries are collected from each patient and filled out on non-consecutive days. Patients are asked to record their urination times, the amount of urine produced, and their activities at the time of any leakage, including the corresponding times.

SECONDARY OUTCOMES:
Pelvic Floor Muscle Strength (PFMS) | 12 WEEKS
  Pelvic Floor Muscle Strength (PFMS) will be evaluated using the digital palpation method, which is a low-cost, easy-to-apply, and widely used reliable assessment tool in clinical practice. In this study, participants will be positioned in the supine position with their knees in flexion and abduction, and a pillow will be placed under their heads. The assessing physiotherapist will insert the index and middle fingers horizontally into the vaginal canal and will ask the participant to contract the pelvic floor muscles as if attempting to stop the flow of urine or gas. The strength of the muscle contraction felt around the fingers will be assessed using the Modified Oxford Scale, a widely used grading system in the literature ranging from 0 to 5. An increase in the score will indicate an improvement in pelvic floor muscle strength.
Quality of Life Assessment | 12 WEEKS
  The King Health Questionnaire (KHQ) will evaluate the patient's quality of life. The KHQ is a commonly used survey comprising 32 items divided into two sections. It is designed to assess patients' quality of life with urinary incontinence. In addition to two single-item questions regarding general health status and quality of life impact, it includes seven subheadings made up of multiple items: role limitations, physical limitations, social limitations, limitations in personal relationships, emotional problems, sleep, and energy disturbances related to urinary incontinence, and severity measurements for urinary incontinence. The second section is the 11-item Symptom Severity Scale, which evaluates the presence and severity of urinary symptoms. The score for the Symptom Severity Scale ranges from 0 (best) to 30 (worst). Scores for other KHQ areas range from 0 (best) to 100 (worst). A higher score indicates a deterioration in the patient's quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Zengin Alpozgen, Assoc. Prof., Principal Investigator — Istanbul University - Cerrahpasa; Aycan Cakmak Reyhan, Asst. Prof., Study Chair — Istanbul Bilgi University
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)